CLINICAL TRIAL: NCT04500899
Title: Evaluating the Severity of Mitral Regurgitation Using Phenylephrine During Transesophageal Echocardiography
Brief Title: Use of Phenylephrine for Assessment of Mitral Regurgitation Severity
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-11414
Record Dates: First submitted 2020-07-23; First posted 2020-08-05 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Oxymetazoline; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mydfrin (Experimental): Phenylephrine is available as phenylephrine hydrochloride injection, 10 mg/mL in 1 mL vial. For intravascular bolus administration, the investigators will prepare a solution containing 100 mcg/mL of phenylephrine hydrochloride, by withdrawing 10 mg (1ml of 10mg/mL) of phenylephrine injection and diluting with 99 mL of 5% dextrose injection or 0.9% sodium chloride injection.
  Interventions: Drug: Mydfrin

INTERVENTIONS:
Drug: Mydfrin — A test dose of 20 mcg of Mydfrin will be administered through the peripheral intravenous line. BP will be monitored after each bolus of phenylephrine. Subsequent Mydfrin injections will then be administered in 50 mcg aliquots every 10-15 minutes, instead of 40 mcg, until the mean arterial blood pressure (MAP) increases by ≥ 20 mm Hg from the baseline MAP, however making sure not to exceed a MAP of 100 mmHg. Once a desired blood pressure has been achieved and maintained, echocardiographic evaluation of mitral regurgitation would be performed.
  Other Names: Phenylephrine

SUMMARY:
The study proposes to develop a phenylephrine protocol to be used during transesophageal echocardiography, whereby intravenous phenylephrine would be used to increase afterload with the intent to mimic the awake hemodynamic profile and variation that occurs with normal physical activity. The expectation is to see changes in severity of Mitral Regurgitation (MR) grade with increasing afterload, which in turn can provide more accurate quantification of MR severity to assist in clinical decision making.

DETAILED DESCRIPTION:
Routine echocardiography which is used to assess the severity of mitral regurgitation, sometimes underestimates the severity of mitral regurgitation, due to hemodynamic variations that occurs with normal physical activity and under the effect of sedation which is used to perform transesophageal echocardiography. By using phenylephrine during transesophageal echocardiography, the study intends to offset the hemodynamic variation that occurs with sedation and better assess the severity of mitral regurgitation, which would further assist in clinical decision-making regarding treatment. The goal of this study is to compare the severity of mitral regurgitation grade before and after the administration of phenylephrine during transesophageal echocardiography and to demonstrate a 25% increase in severity of mitral regurgitation grade compared to the baseline conditions, following the administration of phenylephrine.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with MR on baseline echocardiographic evaluation who are scheduled to undergo TEE for further evaluation of mitral regurgitation.

Exclusion Criteria:

* The following patients will be excluded from the study:

  1. Patients who are not clinically eligible for TEE.
  2. Patients with contraindications to esophageal intubation.
  3. Patients with hemodynamic instability.
  4. Patients with acute decompensated heart failure (HF).
  5. Patients with un-revascularized severe coronary artery disease (triple vessel or left main disease).
  6. Patients with ongoing unstable angina or ongoing myocardial infarction (MI)
  7. Patients with significant arrhythmias including atrial fibrillation.
  8. Patients with uncontrolled hypertension (BP ≥ 150/90 mmHg).
  9. Patients with preexisting bradycardia (HR < 50) and heart blocks.
  10. Patients with severe symptomatic peripheral vascular disease.
  11. Patients with severe pulmonary hypertension (estimated systolic pulmonary arterial pressure sPAP ≥ 60mm Hg).
  12. Patients who are at high risk for intracranial bleeding such as patients with previous strokes, transient ischemic attack (TIA) and vascular malformations.
  13. Additionally, patients with mean arterial blood pressure MAP > 100 mmHg during TEE and those with severe MR, effective regurgitant orifice area (ERO > 39cm2) on baseline TEE evaluation will not be given phenylephrine and excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with greater than 25% increase in MR regurgitant volume (Rvol) after the use of phenylephrine during transesophageal echocardiography. | Before and after phenylephrine administration during transesophageal echocardiography, approximately 40 minutes
  The purpose of this study is to compare the echocardiographic parameters of MR grade before and after the use of phenylephrine during transesophageal echocardiography (TEE) and to document an increase in echocardiographic parameters of MR grade after the use of phenylephrine.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Garcia, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carabello BA. The current therapy for mitral regurgitation. J Am Coll Cardiol. 2008 Jul 29;52(5):319-26. doi: 10.1016/j.jacc.2008.02.084. PMID 18652937
- [Background] Lehmann KG, Francis CK, Dodge HT. Mitral regurgitation in early myocardial infarction. Incidence, clinical detection, and prognostic implications. TIMI Study Group. Ann Intern Med. 1992 Jul 1;117(1):10-7. doi: 10.7326/0003-4819-117-1-10. PMID 1596042
- [Background] Singh JP, Evans JC, Levy D, Larson MG, Freed LA, Fuller DL, Lehman B, Benjamin EJ. Prevalence and clinical determinants of mitral, tricuspid, and aortic regurgitation (the Framingham Heart Study). Am J Cardiol. 1999 Mar 15;83(6):897-902. doi: 10.1016/s0002-9149(98)01064-9. PMID 10190406
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Jul 11;70(2):252-289. doi: 10.1016/j.jacc.2017.03.011. Epub 2017 Mar 15. No abstract available. PMID 28315732
- [Background] Shiran A, Merdler A, Ismir E, Ammar R, Zlotnick AY, Aravot D, Lazarovici H, Zisman E, Pizov R, Lewis BS. Intraoperative transesophageal echocardiography using a quantitative dynamic loading test for the evaluation of ischemic mitral regurgitation. J Am Soc Echocardiogr. 2007 Jun;20(6):690-7. doi: 10.1016/j.echo.2006.11.004. PMID 17543738
- [Background] Sanfilippo F, Johnson C, Bellavia D, Morsolini M, Romano G, Santonocito C, Centineo L, Pastore F, Pilato M, Arcadipane A. Mitral Regurgitation Grading in the Operating Room: A Systematic Review and Meta-analysis Comparing Preoperative and Intraoperative Assessments During Cardiac Surgery. J Cardiothorac Vasc Anesth. 2017 Oct;31(5):1681-1691. doi: 10.1053/j.jvca.2017.02.046. Epub 2017 Feb 13. PMID 28506541
- [Background] Kolev N, Brase R, Wolner E, Zimpfer M. Quantification of mitral regurgitant flow using proximal isovelocity surface area method: a transesophageal echocardiography perioperative study. J Cardiothorac Vasc Anesth. 1998 Feb;12(1):22-6. doi: 10.1016/s1053-0770(98)90050-7. PMID 9509352
- [Background] Recusani F, Bargiggia GS, Yoganathan AP, Raisaro A, Valdes-Cruz LM, Sung HW, Bertucci C, Gallati M, Moises VA, Simpson IA, et al. A new method for quantification of regurgitant flow rate using color Doppler flow imaging of the flow convergence region proximal to a discrete orifice. An in vitro study. Circulation. 1991 Feb;83(2):594-604. doi: 10.1161/01.cir.83.2.594. PMID 1991377